CLINICAL TRIAL: NCT04552717
Title: My Grief - Development and Evaluation of an App for Parents With Prolonged Grief Disorder After Losing a Child to Cancer: a Randomized Controlled Trial
Brief Title: My Grief - an App for Parents With Prolonged Grief After Losing a Child to Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Josefin Sveen, PhD, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-01704
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Prolonged Grief Disorder
MeSH Terms: conditions — Prolonged Grief Disorder

STUDY DESIGN:
Intervention Model Description: wait-list controll and intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will complete a web based pre-assessment and then given access to the app "My Grief" for three months followed by a web based post-assessment and an interview via telephone regarding their experiences of using the app, and follow-up questionnaires.
  Interventions: Other: My Grief
- Waitlist controll (No Intervention): Participants will get access to the app after three months.

INTERVENTIONS:
Other: My Grief — The app will build on principles of cognitive behavioural theory and therapy (CBT) and contains four main sections: Learning, Self-assessment, Manage symptoms and Find support.
  Arms: Intervention

SUMMARY:
Bereaved parents are at increased risk of developing mental and physical health problems and bereavement is even associated with an increased risk of mortality, especially in mothers. Prolonged grief disorder (PGD) are persistent and intensive grief reactions which can persist for years. It is characterized by an intense and lasting yearning for the deceased, intense emotional pain, such as difficulty accepting the loss and an inability to experience positive mood. Parents are among the most vulnerable to develop PGD.

The goal is to increase the accessibility to evidence-based and cost-effective interventions for parents of children who have died of cancer, and thus facilitate the grieving process and decrease the risk for parents to develop long-term distress.

Specific aims are:

* To evaluate the acceptability and feasibility of a mobile app, "My Grief ", a self-help app for prolonged grief, in parents who lost a child to cancer.
* To evaluate possible beneficial effects of the mobile app on parents' mental health.

DETAILED DESCRIPTION:
There is a lack of studies evaluating the effect of interventions for bereaved parents. Thus, there is a need for accessible interventions with documented efficacy for preventing or reducing negative mental health consequences after the loss of a child. Today, many individuals carry smartphones and these devices can be used to access self-help interventions aiming to improve both physical and mental health. Currently, there are an excess of apps available for smartphone users that assert that they help people with their physical or mental health. However, for most of these apps, there is a lack of empirical support, i.e., their efficacy is unknown. It is therefore important to evaluate mobile apps in scientific studies with rigorous designs. In addition, before conducting rigorous studies of novel psychosocial interventions, such as a mobile app, it is important to conduct more basic work evaluating development and feasibility of the intervention. One such self-help app, the PTSD Coach, has been evaluated in a randomized controlled trial conducted with traumatized participants recruited from the community, which found that access to the PTSD Coach app was associated with improvements in posttraumatic stress (PTS) symptoms, depression, and psychosocial functioning. The PTSD Coach app is based on cognitive behavioural therapy (CBT) principles and there is a growing body of evidence that elements of CBT are effective interventions for prolonged grief. Thus, an app targeting prolonged grief using elements of CBT could potentially be effective in improving the mental health in bereaved parents. To our knowledge no such app has been developed and evaluated. The Grief Coach app will be based on the smartphone app PTSD Coach. A Swedish version of the PTSD Coach has been developed and a pilot study has been conducted as well as an ongoing RCT. Consultant programmers at Uppsala University will develop the mobile app. The content of the app will be developed together with experts in the field of grief, inspired by other grief apps and CBT therapy manuals, to modify parts of the PTSD Coach app to grief.

The main aim of this study is to examine the effectiveness of the app My Grief as compared to a waiting list comparison in reducing symptoms of prolonged grief in bereaved parents. The primary hypothesis is that the parents in the intervention group will report decreased levels of prolonged grief symptoms after having used the app. A second aim is to examine the effect of the app on related mental health problems (posttraumatic stress symptoms, depression symptoms, quality of life) and cognitive behavioral variables putatively explaining the effect of CBT techniques (i.e., grief avoidance, grief rumination and negative grief cognitions). The secondary hypotheses are that the parents in the intervention group will report improved mental health (i.e., lower symptom levels of depression and posttraumatic stress, higher quality of life), and lower grief avoidance, grief rumination, negative grief-related cognitions. A third aim is to evaluate the feasibility of the app, including participant satisfaction, evaluation of the app's strengths and weaknesses, and adverse events.

Potential participants are identified using the Swedish Childhood Cancer Registry, the Cause of Death Registry, and the Swedish Population Register at the Swedish Tax Agency. By linking the Cause of Death Registry with the Swedish Childhood Cancer Registry, children diagnosed with a malignancy and who died due to the malignancy 1 to 10 years previously will be identified. Next, the children's parents/caregivers are identified through the Swedish Population Register and will be sent a letter with an invitation to participate in the study. Participants will complete a web based pre-assessment and then given access to the app for three months followed by a web based post-assessment and an interview via telephone regarding their experiences of using the app, with follow-ups att 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers of children who have died of cancer, at the earliest 12 month ago
* Have symptoms of prolonged grief (PGD)
* Understand Swedish language
* Have access to a smartphone

Exclusion Criteria:

* Ongoing severe psychiatric problems (e.g. suicidal thoughts, psychosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Change (from baseline) in Prolonged Grief Disorder-13 instrument, PG-13 | 3, 6 and 12 months
  13-item, self-rated measure of prolonged grief, total score ranges from 11 to 55, where a higher score indicates more symptoms

SECONDARY OUTCOMES:
Change (from baseline) in Posttraumatic stress disorder checklist for DSM-5, PCL-5 | 3, 6 and 12 months
  20-item, self-rated measure of posttraumatic stress disorder, total score range from 0-80, and a higher score indicates more symptoms
Change (from baseline) in Patient Health Questionnaire, PHQ-9 | 3, 6 and 12 months
  9-item, self-rated measure of depression, total score ranges from 0-27, and a higher score indicates more symptoms
Change (from baseline) in Utrecht Grief Rumination Scale, UGRS | 3, 6 and 12 months
  15-item, self-rated measure of grief rumination, total scores range from 15 to 75, and a higher score indicates more grief rumination
Change (from baseline) in Depressive and Anxious Avoidance in Prolonged Grief questionnaire | 3, 6 and 12 months
  9-item, self-rated measure of avoidance, total score ranges from 9-72, and a higher score indicates more avoidance
Change (from baseline) in 18 items from the Grief Cognitions Questionniare, GCQ | 3, 6 and 12 months
  18-items, self-rated measure of grief cognitions, total score ranges from 0-90, and a higher score indicates more grief cognitions
Change (from baseline) in Brunnsviken Brief Quality of Life Inventory, BBQ | 3, 6 and 12 months
  12 items, self-rated measure of quality of life, covering six different life domains, Total score ranges from 0-96, higher scores indicates higher quality of life.

OTHER OUTCOMES:
Feasibility of the intervention and the application | 3 months
  Feasibility will be measured by "App Survey"
Acceptability of the intervention and the application | 3 months
  Acceptability will be measured by "App Survey"
Participants demographics | 0 months
  age, gender, time since loss, gender child, marital status, employment status, loss-related variables

CONTACTS AND LOCATIONS:
Overall Officials: Josefin Sveen, PhD, Principal Investigator — Uppsala University
Locations (1):
- National Centre for Disaster Psychiatry, Department of Neuroscience, Uppsala university, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Sveen J, Eisma MC, Boelen PA, Arnberg FK, Eklund R. My grief app for prolonged grief in bereaved parents: a randomised waitlist-controlled trial. Cogn Behav Ther. 2025 Jul;54(4):514-530. doi: 10.1080/16506073.2024.2429068. Epub 2024 Nov 14. PMID 39540459
- [Derived] Eklund R, Eisma MC, Boelen PA, Arnberg FK, Sveen J. My Grief App for Prolonged Grief in Bereaved Parents: A Pilot Study. Front Psychiatry. 2022 Apr 25;13:872314. doi: 10.3389/fpsyt.2022.872314. eCollection 2022. PMID 35546953
- [Derived] Eklund R, Eisma MC, Boelen PA, Arnberg FK, Sveen J. Mobile app for prolonged grief among bereaved parents: study protocol for a randomised controlled trial. BMJ Open. 2021 Dec 7;11(12):e052763. doi: 10.1136/bmjopen-2021-052763. PMID 34876429